CLINICAL TRIAL: NCT00260416
Title: Primary Angioplasty for Acute Myocardial Infarction in Patients With Symptom Duration Above 12 Hours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Danish Heart Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STEMI-12
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Symptom duration; Primary angioplasty; Infarct size; Myocardial scintigraphy
MeSH Terms: interventions — Stents; Abciximab

INTERVENTIONS:
Procedure: Primary angioplasty with stent and abciximab

SUMMARY:
Background: Acute balloon angioplasty is beneficial in patients with acute myocardial infarction. However, presently this treatment is not offered to patients with symptom duration above 12 hours.

Hypothesis: Acute balloon angioplasty for myocardial infarction is beneficial despite symptom duration above 12 hours.

Methods: In 60 patients with myocardial infarction and symptom duration above 12 hours, the proportion of non-perfused myocardium before acute angioplasty and 1 month after angioplasty is compared to evaluate if myocardial tissue can be saved by acute angioplasty despite long symptom duration.

DETAILED DESCRIPTION:
Methods: On arrival at our angioplasty laboratory, patients are informed about the study. If they accept to participate, we infuse 600 MBq of Sestamibi i.v. This binds in a first passage fashion without later redistribution to perfused myocardium. Non-perfused myocardium does not bind sestamibi. Primary angioplasty with stent and abciximab is then performed followed by myocardial scintigraphy to illustrate the non-perfused myocardial area that was at risk of infarction before the coronary artery was opened. Echocardiography is also performed. At 1 month, myocardial scintigraphy is repeated to evaluate infarct size. The difference between the myocardial area at risk of infarction before angioplasty and the myocardial infarct size 1 month later is defined as "salvage". Scintigraphy is repeated at 6 month and echocardiography is also repeated at 1 month and 6 months. The primary endpoint is "salvage". Accordingly, the aim is to demonstrate that salvage can be achieved with primary angioplasty for acute myocardial infarction despite symptom duration above 12 hours. Clinical endpoints are death and reinfarction. The results are compared with results in 200 patients with symptom duration below 12 hours. These patients are treated and examined according to the exact same protocol. By this comparison, it can be evaluated whether it is relevant that the current guidelines recommend acute balloon angioplasty only to patients with less than 12 hours of symptom duration.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction with ST-segment elevation;
* Symptom duration 12 hours to 72 hours.

Exclusion Criteria:

* Age below 18 years;
* Bleeding disorders or anaemia or low levels of thrombocytes;
* Thrombolysis used during the present admission;
* Expected survival less than 1 year due to other diseases;
* Previous acute myocardial infarction or coronary by-pass surgery;
* Major operation within last 30 days;
* Heamorrhaghic stroke within last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Myocardial salvage as evaluated by repeat myocardial scintigraphy(= area at risk of infarction before primary angioplasty - infarct size at 1 month).

SECONDARY OUTCOMES:
Infarct size by myocardial scintigraphy at 1 month and 6 months after primary angioplasty.
Death at 1 month and 6 months.
Reinfarction at 1 month and 6 months.
Ejection fraction at 1 day, 1 month and 6 months.
Left ventricular end diastolic volume at 1 day, 1 month and 6 months.
Brain Natriuretic Peptide levels at 1 day, 1 month and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Steen D. Kristensen, MD, Study Director — Dept. of Cardiology, Skejby Hospital, AarhusUniversity Hospital, DK-8200 Aarhus N, Denmark, Europe
Locations (1):
- Departments of Cardiology and Nuclear Medicine at Skejby Hospital, Aarhus, Denmark